CLINICAL TRIAL: NCT00888498
Title: Ankle Manual Therapy for Individuals With Post-Acute Ankle Sprains: A Randomized, Placebo-Controlled Trial
Brief Title: Ankle Manual Therapy for Ankle Sprains
Acronym: AMT
Status: Suspended | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of the Pacific (Other)
Collaborators: University of Southern California (Other); American Physical Therapy Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UPacific
Record Dates: First submitted 2009-04-24; First posted 2009-04-27 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-07

CONDITIONS: Sprains and Strains
Keywords: Sprains and Strains; Ankle; Manual Therapies; Outcome Studies
MeSH Terms: conditions — Sprains and Strains | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Hands-On Control (Placebo Comparator): With the subject in a seated position on a treatment table and the lower extremity of interest stabilized to the table with a belt, a single standardized treating investigator will grasp the foot of interested with the thenar eminences on the foot's plantar surface, which is similar to the positioning used for the experimental groups. The treating investigator will maintain passive positioning of the ankle for the duration of 1 deep inhalation and exhalation by the subject rather than induce an iatrogenic force.
  Interventions: Other: Passive Positioning
- Fast Stretching (Experimental): With the subject in a seated position on a treatment table and the lower extremity of interest stabilized to the table with a belt, a single standardized treating investigator will grasp the foot of interested with the thenar eminences on the foot's plantar surface. A thrust will be delivered parallel to the long axis of the subject's lower leg after the treating therapist induces passive ankle dorsiflexion to end range.
  Interventions: Other: High-Velocity, Low-Amplitude Stretch
- Slow Stretching (Experimental): With the subject in a seated position on a treatment table and the lower extremity of interest stabilized to the table with a belt, a single standardized treating investigator will grasp the foot of interested with the thenar eminences on the foot's plantar surface. Traction will be delivered to the talocrural joint at the treating therapist's second perception of tissue resistance in 3 bouts of 30-second holds, separated by 10 seconds of rest.
  Interventions: Other: Slow, Mobilization Stretch

INTERVENTIONS:
Other: Passive Positioning — With the subject in a seated position on a treatment table and the lower extremity of interest stabilized to the table with a belt, a single standardized treating investigator will grasp the foot of interested with the thenar eminences on the foot's plantar surface, which is similar to the positioning used for the active comparator groups. The treating investigator will maintain passive positioning of the ankle for the duration of 1 deep inhalation and exhalation by the subject rather than induce an iatrogenic force.
  Other Names: Manual Therapy
  Arms: Hands-On Control
Other: High-Velocity, Low-Amplitude Stretch — With the subject in a seated position on a treatment table and the lower extremity of interest stabilized to the table with a belt, a single standardized treating investigator will grasp the foot of interested with the thenar eminences on the foot's plantar surface. A thrust will be delivered parallel to the long axis of the subject's lower leg after the treating therapist induces passive ankle dorsiflexion to end range.
  Other Names: Manual Therapy
  Arms: Fast Stretching
Other: Slow, Mobilization Stretch — With the subject in a seated position on a treatment table and the lower extremity of interest stabilized to the table with a belt, a single standardized treating investigator will grasp the foot of interested with the thenar eminences on the foot's plantar surface. Traction will be delivered to the talocrural joint at the treating therapist's second perception of tissue resistance in 3 bouts of 30-second holds, separated by 10 seconds of rest.
  Other Names: Manual Therapy
  Arms: Slow Stretching

SUMMARY:
The purpose of this study is to determine the effect of using ankle manual therapy procedures on clinical outcomes in individuals with post-acute ankle sprains.

DETAILED DESCRIPTION:
Ankle sprains can cause ankle joint stiffness. Ankle joint stiffness may be a cause of pain, disability, and repeated sprains. Physical therapists use many ways to treat ankle joints that do not move well. One way takes 1-2 seconds. Another way may take up to 1 minute. Both kinds of stretches seem to improve ankle flexibility. However, we do not know how well they work to improve pain and disability in individuals following ankle sprains. The purpose of this research is to find out which physical therapy treatments work best for people with ankle sprains. To start the study, subjects will be asked to fill out some forms that ask about their ankle problem. Subjects will receive an examination by a physical therapist that includes gentle movements of the feet and legs to test their flexibility, strength, and balance. Subjects will then be assigned to 1 of 3 treatments to be provided by a separate physical therapist. They will not get to choose their group. All 3 groups will receive ankle stretching by the physical therapist. The groups will differ in how much and how fast the stretch will be. The first group will have an ankle stretch that lasts 1-2 seconds. The second group will have a stretch that lasts 1 minute. The third group will have their foot held without any stretching. After stretching, all subjects will receive the same kind of exercise program. Study-related treatment will last 5 sessions over 4 weeks, with 2 sessions for stretching within the 1st week and 1 session per week for the 3 following weeks for the exercise program. After 1 week and 4 weeks, subjects will fill out the same forms as at the initial examination. The treatment part of the study will then be finished. After 6 months, 1 year, and 2 years from enrollment in the study, subjects be asked to fill out many of the same forms that ask about their ankle problem. We think subjects that get a stretch will have a better outcome than subjects that get ankle holding. To test our idea, we will compare how subjects in each group tell us they are doing with their ankle problem on the Foot and Ankle Ability Measure at 1 week, 4 weeks, 6 months, 1 year, and 2 years following entry into the study. Since the way a person thinks and feels about their injury may have something to do with how much they improve during physical therapy, we will also measure these factors to find out if they affect the results of this study.

ELIGIBILITY:
Inclusion Criteria:

* Age 16-60 years
* Onset of ankle sprain at least 2 weeks prior to enrollment
* Foot and Ankle Ability Measure Activity of Daily Living subscale score less than or equal to 80%

Exclusion Criteria:

* Current status of assisted ambulation (eg, use of cane or crutches)
* Inability to bear weight through the affected extremity immediately after injury combined with tenderness to palpation of the medial and lateral malleolar zones, styloid process of the 5th metatarsal, and navicular
* Positive anterior drawer or talar tilt dimple test
* Volume of the affected limb greater than 10% of the unaffected limb
* Previous history of ligament or bony reconstructive surgery to the ankle and foot
* Concomitant injury to other lower extremity joints

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 189 (Estimated)
Dates: Start 2009-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Foot and Ankle Ability Measure | Intake, 1 week, 4 weeks, 6 months, 1 year, 2 years

SECONDARY OUTCOMES:
Patient Global Rating of Improvement | Intake, 1 week, 4 weeks, 6 months, 1 year, 2 years
Modified Fear Avoidance Beliefs Questionnaire | Intake, 1 week, 4 weeks, 6 months, 1 year, 2 years
Lower Extremity Self Efficacy Scale | Intake, 1 week, 4 weeks, 6 months, 1 year, 2 years
Positive and Negative Affect Scale | Intake, 1 week, 4 weeks, 6 months, 1 year, 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Todd E Davenport, PT, DPT, OCS, Principal Investigator — University of the Pacific; Kornelia Kulig, PhD, PT, Study Director — University of Southern California; Beth Fisher, PhD, PT, Study Director — University of Southern California
Locations (1):
- University of the Pacific, Stockton, California, United States

REFERENCES:
- [Derived] Davenport TE, Kulig K, Fisher BE. Ankle manual therapy for individuals with post-acute ankle sprains: description of a randomized, placebo-controlled clinical trial. BMC Complement Altern Med. 2010 Oct 19;10:59. doi: 10.1186/1472-6882-10-59. PMID 20958995